CLINICAL TRIAL: NCT06575881
Title: Defining the Risk of Ventricular Tachycardia in Genetic Forms of Early-onset Atrial Fibrillation
Brief Title: Defining the Risk of Ventricular Tachycardia in Genetic Cardiomyopathies
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, M. Benjamin Shoemaker, Associate Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: IRB231260
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Ventricular Tachycardia; Premature Ventricular Contraction
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular; Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TTN-positive: Patients with a pathogenic or likely pathogenic variant in TTN on clinical genetic testing.
- Gene-positive: Patients with a pathogenic or likely pathogenic variant in a gene other than TTN on clinical genetic testing.
- Gene-negative: Patients without a pathogenic or likely pathogenic variant in a cardiomyopathy or arrhythmia gene on clinical genetic testing.

SUMMARY:
The goal of this observational study is to determine if electrophysiologic mapping and cardiac MRI can help identify patients that have genetic forms of cardiomyopathy that are at high risk for development of dangerous ventricular arrhythmias.

The investigators aim to study:

1. the prevalence and mechanism of inducible ventricular tachycardia
2. pace-mapping to define the site of origin of ventricular arrhythmias
3. voltage mapping to define low voltage scar substrate in the basal LV to determine the risk of development of ventricular arrhythmias in patients with genetic forms of cardiomyopathy.

Participants will undergo cardiac MRI before their scheduled procedure and voltage mapping during their scheduled procedure as part of data collection.

DETAILED DESCRIPTION:
New genomic knowledge is poised to change clinical practice for atrial fibrillation (AF). In 1293 cases previously considered idiopathic, the investigators identified a pathogenic variant in a cardiomyopathy (CM) or arrhythmia gene in ~11% of patients diagnosed with AF before age 608 and went on to show that these patients have a higher risk of mortality and sudden death. The investigators propose tests of specific hypotheses that will address the major knowledge gap of whether and how genetic findings should change clinical management recommendations.

Aim: To use programmed ventricular stimulation at the time of AF ablation or Electrophysiology Study to define the prevalence and mechanism of inducible ventricular tachycardia (VT) (Aim 1A); pace-mapping to define the site of origin of ventricular arrhythmias (Aim 1B); and voltage mapping to define low voltage scar substrate in the basal LV (Aim 1C) in patients with pathogenic TTN variants compared to genotype-negative controls.

The Aim is informed by the observation that life-threatening VT in patients with dilated CM and pathogenic TTN variants most often localizes to the LV outflow tract (LVOT), periaortic region, and basal septum. The investigators found that 39% (27/70) of patients with early-onset AF and pathogenic TTN variants have premature ventricular contractions (PVCs) and non-sustained VT that localize to this same area, which the investigators therefore hypothesize are an early marker of a malignant arrhythmia substrate. Life-threatening ventricular arrhythmias are usually due to scar-related reentry, but a major problem with the LVOT/periaortic region is that scar in this area is hard to detect. To address this limitation, the investigators have published new voltage cutoffs to define scar in the LVOT/periaortic region. The Aim addresses the overarching hypothesis that patients with pathogenic TTN variants have occult scar in the basal LV and are at risk for life-threatening reentrant VT. The investigators will define the mechanism of VT using a combination of entrainment maneuvers with overdrive pacing and the identification of scar with voltage mapping. To facilitate the Aim, the investigators have established a dedicated AF Precision Medicine Clinic to evaluate patients with early onset AF. Fifty percent of these patients undergo AF ablation for symptomatic AF, which the investigators have found is as effective in TTN patients as genotype-negative controls. The investigators will enroll 50 patients with a pathogenic variant in TTN, 50 with a pathogenic variant in other CM genes (e.g., LMNA), and 100 genotype-negative controls.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Diagnosed with AF, frequent PVCs, or VT before age 60
* Scheduled for catheter-based AF ablation (de-novo or repeat) OR catheter-based PVC ablation OR catheter-based VT ablation
* Able to provide written, informed consent
* P/LP variant in TTN or other CM gene (cases) or identified as a genotype-negative control.

Exclusion Criteria:

* Diagnosed with a genetic CM or arrhythmia syndrome prior to ablation procedure
* VUS in 'possibly pathogenic' subgroup (control group only)
* Previous PVC or VT ablation
* LVEF <20%
* Prosthetic mitral or aortic valve
* Contraindication to heparin
* Prior myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Young patients with atrial fibrillation, frequent PVCs, or VT that are scheduled to undergo procedural management of their arrhythmia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Ventricular Tachycardia Inducibility | During procedure
  Patients will undergo an electrophysiology study (EP study) as part of the research or clinical protocol for the procedure. Inducible VT (yes/no) with the EP study will be the primary outcome measure.

SECONDARY OUTCOMES:
Site and Substrate of Ventricular Ectopy | During procedure
  Localization of ventricular ectopy or arrhythmia will be evaluated during the procedure by electoanatomic mapping, and the assessment of scar burden in this area (by voltage mapping) will be secondary outcomes for Aims 1B and 1C.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States